CLINICAL TRIAL: NCT06009523
Title: Effects of Transcranial Direct Current Stimulation (tDCS) in the Management of Suicidal Ideation in Treatment-resistant Depression : a Pilot Study
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) in the Management of Suicidal Ideation
Acronym: tDCS-IDSDEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01454-39
Record Dates: First submitted 2023-08-01; First posted 2023-08-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression and Suicide
Keywords: tDCS
MeSH Terms: conditions — Depression; Suicide | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active tDCS (Experimental): Participants received an active tdcs: transcranial direct current with an intensity of 2 mA for 30 minutes
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — 1 stimulation per day during 15 days.

SUMMARY:
The main objective of this study is to demonstrate that 15 transcranial direct current stimulation (tDCS) sessions of 30 minutes at 2 mA intensity are effective to reduce suicidal ideation

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening visit to determine eligibility for study entry. Patient who meet the eligibility requirements be able to start the 15 tDCS sessions at the rate of one session per day. After the last session, patients will perform three follow-up visits on D19, D49 and D79

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Written informed consent
* Diagnosis of recurrent or isolated depressive episode according to DSM IV criteria (A.P.A. 1994).
* Stable antidepressant treatment for 3 weeks
* MADRS score ≥ 20
* SSI score > 3
* Subject affiliated to a health insurance system
* Woman with effective contraception and agreeing to maintain it throughout the study period.

Exclusion Criteria:

* Depression with psychotic features Axis I (DSM IV) co-morbid diagnosis of schizophrenia, alcohol and/or other substance dependence (or abuse) (lifetime)
* Patient who has already undergone an electroconvulsive therapy course for the current episode and does not respond to this treatment
* Patient deprived of liberty
* Patient with high suicide risk (item 10 MADRS > 4) in the absence of hospitalization
* Contraindication to tDCS: intracerebral metallic implant (with the exception of dental implants), cardiac pacemaker, active or non-implanted devices in the region of the head, acute eczema in the planned stimulation area
* Pregnant, parturient or breastfeeding woman
* Simultaneous participation in another interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in suicidal ideation on the Scale for Suicide Ideation (SSI) at "Day 19" | Baseline and "Day 19"
  The main judgment criterion is the evolution of suicidal ideation which is evaluated by the Beck Scale for Suicide Ideation (SSI) between Baseline and "Day 19"

SECONDARY OUTCOMES:
Change from Baseline of clinical response defined by the MADRS (Montgomery and Asberg depression scale) at "Day 19" post-tDCS sessions | Baseline and "Day 19"
  The Montgomery-Åsberg Depression Rating Scale (MADRS) was developed to provide an assay of depressive symptom severity for use in the investigation of treatment response to antidepressant medication. The MADRS takes 20-60 minutes to be completed by interview. MADRS-S has 9 items , and each item is scored between 0 (minimum) and 6 (maximum). The scores for all 9 items were added, and cutoff scores for the MADRS-S were defined for level of depression (depression: 0-12 = minimal, 13-19 = mild, 20-34 = moderate, ≥ 35 = severe).
Change from Baseline of clinical response defined by the MADRS (Montgomery and Asberg depression scale) at "Day 49" post-tDCS sessions | Baseline and "Day 49"
  The Montgomery-Åsberg Depression Rating Scale (MADRS) was developed to provide an assay of depressive symptom severity for use in the investigation of treatment response to antidepressant medication. The MADRS takes 20-60 minutes to be completed by interview. MADRS-S has 9 items , and each item is scored between 0 (minimum) and 6 (maximum). The scores for all 9 items were added, and cutoff scores for the MADRS-S were defined for level of depression (depression: 0-12 = minimal, 13-19 = mild, 20-34 = moderate, ≥ 35 = severe).
Change from Baseline of clinical response defined by the MADRS (Montgomery and Asberg depression scale) at "Day 79" post-tDCS sessions | Baseline and "Day 79"
  The Montgomery-Åsberg Depression Rating Scale (MADRS) was developed to provide an assay of depressive symptom severity for use in the investigation of treatment response to antidepressant medication. The MADRS takes 20-60 minutes to be completed by interview. MADRS-S has 9 items , and each item is scored between 0 (minimum) and 6 (maximum). The scores for all 9 items were added, and cutoff scores for the MADRS-S were defined for level of depression (depression: 0-12 = minimal, 13-19 = mild, 20-34 = moderate, ≥ 35 = severe).
Change from Baseline in suicidal ideation assessed by the implicit association test at "Day 19" post-tDCS sessions | Baseline and "Day 19"
  The Implicit Association Test (IAT) is a computer-based test measuring implicit mental associations between two concepts. The IAT uses reaction times to categorize stimuli that appear in the middle of the screen into two target categories, in our study: "Death" (suicide, dies, funeral, lifeless, deceased) and "Life". (survive, grow, breathe, alive, live) and/or in two attribute categories "Me" (me, myself, my, mine, I) and "Not Me" (them, they, their, his, others) . and subjects rapidly classify them by pressing one of two keys (the category of right (by pressing the I key) or left (by pressing the E key). According to the logic of the IAT, "D positive" scores represent a strong implicit association between "Me" and "Death". We will use Greenwald's improved algorithm to analyze responses.
Change from Baseline in suicidal ideation assessed by the implicit association test at "Day 49" post-tDCS sessions | Baseline and "Day 49"
  The Implicit Association Test (IAT) is a computer-based test measuring implicit mental associations between two concepts. The IAT uses reaction times to categorize stimuli that appear in the middle of the screen into two target categories, in our study: "Death" (suicide, dies, funeral, lifeless, deceased) and "Life". (survive, grow, breathe, alive, live) and/or in two attribute categories "Me" (me, myself, my, mine, I) and "Not Me" (them, they, their, his, others) . and subjects rapidly classify them by pressing one of two keys (the category of right (by pressing the I key) or left (by pressing the E key). According to the logic of the IAT, "D positive" scores represent a strong implicit association between "Me" and "Death". We will use Greenwald's improved algorithm to analyze responses.
Change from Baseline in suicidal ideation assessed by the implicit association test at "Day 79" post-tDCS sessions | Baseline and "Day 79"
  The Implicit Association Test (IAT) is a computer-based test measuring implicit mental associations between two concepts. The IAT uses reaction times to categorize stimuli that appear in the middle of the screen into two target categories, in our study: "Death" (suicide, dies, funeral, lifeless, deceased) and "Life". (survive, grow, breathe, alive, live) and/or in two attribute categories "Me" (me, myself, my, mine, I) and "Not Me" (them, they, their, his, others) . and subjects rapidly classify them by pressing one of two keys (the category of right (by pressing the I key) or left (by pressing the E key). According to the logic of the IAT, "D positive" scores represent a strong implicit association between "Me" and "Death". We will use Greenwald's improved algorithm to analyze responses.
Change from Baseline in quality-of-life assessed by the SF36 (Short Form (36) Health Survey) at "Day 19" post-tDCS sessions | Baseline and "Day 19"
  The Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is an indicator of overall health status. The SF-36 is validated and has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100, so that the lowest and highest possible scores are 0 and 100, respectively. Lower scores = more disability, higher scores = less disability. Sections : vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Change from Baseline in quality-of-life assessed by the SF36 (Short Form (36) Health Survey) at "Day 49" post-tDCS sessions | Baseline and "Day 49"
  The Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is an indicator of overall health status. The SF-36 is validated and has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100, so that the lowest and highest possible scores are 0 and 100, respectively. Lower scores = more disability, higher scores = less disability. Sections : vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Change from Baseline in quality-of-life assessed by the SF36 (Short Form (36) Health Survey) at "Day 79" post-tDCS sessions | Baseline and "Day 79"
  The Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is an indicator of overall health status. The SF-36 is validated and has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100, so that the lowest and highest possible scores are 0 and 100, respectively. Lower scores = more disability, higher scores = less disability. Sections : vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Nord-Deux-Sèvres, Faye-l'Abbesse
  - Centre Hospitalier Henri Laborit, Poitiers